CLINICAL TRIAL: NCT03846661
Title: Nationwide Long-term Outcome Surveillance of Physiomesh® vs. Other Meshes in Laparoscopic Incisional Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Frederik Helgstrand, Principal Investigator, Zealand University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FH115
Record Dates: First submitted 2019-02-04; First posted 2019-02-20 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Hernia, Abdominal; Recurrence; Postoperative Complications
MeSH Terms: conditions — Hernia, Abdominal; Recurrence; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Register study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physiomesh (Active Comparator): Patients undergoing laparoscopic incisional hernia repair reinforced with a Physiomesh.
  Interventions: Device: Physiomesh
- other mesh (No Intervention): Patients undergoing laparoscopic incisional hernia repair reinforced with other meshes than Physiomesh.

INTERVENTIONS:
Device: Physiomesh — difference in risk for recurrence and postoperative complication
  Other Names: other mesh
  Arms: Physiomesh

SUMMARY:
The primary aim of the present study was to show how a national clinical register combined with other nationwide administrative registers may serve as a tool for pre- and post-marketing evaluation of new mesh and mesh fixation products for hernia surgery, using Physiomesh® versus other meshes designed for laparoscopic hernia repair as an example.

DETAILED DESCRIPTION:
All adult (≥18 yrs) patients registered in the Danish Hernia Database (DHB) who underwent elective primary laparoscopic incisional hernia repair between January 1st 2010 and December 31st 2016.

To obtain 100% follow-up data from DHB will be combined with administrative data from the Danish National Patient register.

Patients will be followed from initial hernia repair until reoperation for recurrence, death, emigration outside Denmark or end of follow-up (november 2017).

Physiomesh and other mesh repairs will be propensity score matched. Each patient in the Physiomesh® group will be matched with two patients treated with one of the other synthetic meshes. The Propensity score includes age, sex, year of surgery, diagnosis of chronic obstructive pulmonary disease, diagnosis of diabetes, diagnosis of obesity, Charlson comorbidity index and size of hernia defect

The primary outcome: Difference in risk for a reoperation for recurrence between patients operated with Physiomesh® and patients operated with another synthetic mesh designed for laparoscopic repair.

The secondary outcome will be rates of 30-day readmission, 30-day reoperation for complications (excluding hernia recurrence) as well as 30- and 90-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients registered in the Danish Hernia Database for a laparoscopic incisional hernia repair

Exclusion Criteria:

* If not registered for a laparoscopic incisional hernia repair in the Danish Hernia Database

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3338 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Re-operation for recurrence rate | up to 84 months

SECONDARY OUTCOMES:
30-day readmission rate | 30 day
30-reoperation for complication rate | 30 day

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Helgstrand, MD, Principal Investigator — Dept. Surgery, Zealand university Hospital
Locations (1):
- Dept. of surgery, Zealand University Hospital, Køge, Denmark